CLINICAL TRIAL: NCT03766321
Title: Interplay Between Gut Microbiota and Adaptive Immunity in Amyotrophic Lateral Sclerosis: a Clinical Trial
Brief Title: Fecal Microbiota Transplantation Effect on Amyotrophic Lateral Sclerosis Patients
Acronym: FETR-ALS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Catholic University of the Sacred Heart (Other); Campus Bio-Medico University (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda Ospedaliera di Perugia (Other); University of Chieti (Other); University of Florence (Other)
Responsible Party: Principal Investigator, JESSICA MANDRIOLI, sponsor-investigator, Azienda Ospedaliero-Universitaria di Modena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FeTr-ALS
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: microbiota; fecal transplantation; adaptive immunity; T regulatory lymphocytes
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: randomized double blind multicentre study on FMT in ALS, with a randomization ratio 2:1 (FMT: placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo will be unrecognizable from active treatment because the patients will undergo endoscopic procedure with sedation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota transplantation (FMT) (Active Comparator): Fecal microbiota transplantation will be performed during two endoscopic procedures (at baseline and at 6 months) by allogenic infusion of collected feces in the duodenum-jejunum. Fecal microbiota will be diluted in saline solution 200 ml and infused at 30 ml/minute speed. Every endoscopic procedure will be performed with sedation of the patient.
  Feces for FMT will be obtained by known healthy donors for C. difficile infection according to standard selection procedures.
  Interventions: Biological: Fecal microbiota transplantation
- Placebo (Placebo Comparator): ALS patients will undergo upper GI endoscopy with small-intestine biopsies at baseline and after 6 months. Patients in the placebo arm will not receive any treatment during these procedures, but will undergo intestinal biopsy.
  Every endoscopic procedure will be performed with sedation of the patient.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fecal microbiota transplantation — Fecal microbiota transplantation will be performed during two endoscopic procedures (baseline and at 6 months) by allogenic infusion of collected feces in the duodenum-jejunum.
  Other Names: FMT
  Arms: Fecal microbiota transplantation (FMT)
Biological: Placebo — patients will undergo endoscopic procedure with biopsy during sedation but without any kind of intervention
  Arms: Placebo

SUMMARY:
Given the role of adaptive immunity in ALS, the pathogenicity of some clostridial strains on motorneurons, the putative role of cyanobacteria in ALS development, and the increasing interest for microbiota in neurodegenerative disorders, the modification of intestinal microbiota might affect ALS at its core.

This interventional study aims at evaluating the biological and disease-modifying effects of Fecal Microbiota Transplant (FMT) in patients affected by Amyotrophic Lateral Sclerosis. As a primary aim of the study, the investigators postulate ALS patients treated with FMT compared to the control arm will display increased Tregs number, which is a favourable biomarker of disease activity and progression. Clinical outcomes as disease progression measured by ALS Functional Rating Scale Revised (ALSFRS-R) score, survival, respiratory function and quality of life will be assessed during the whole treatment and follow-up period.

Moreover, biological activity of FMT will be evaluated in different biomatrices, together with FMT safety and tolerability in a cohort of ALS patients.

DETAILED DESCRIPTION:
The study will include 42 ALS patients with 2:1 allocation in 2 groups of subjects (28 FMT vs 14 placebo); computerized randomization will be stratified by progression rate (ΔFS) </≥0.7. Randomization time will last 18 months. Treatment will be double blinded to patients and physicians, and will be done at baseline and at month 6. FMT is regarded as the active treatment. Post-treatment follow up will be 6 months.

ALS patients will undergo upper GI endoscopy with small-intestine biopsies (n° 4 biopsies of small intestine, performed with a standard biopsy forces) at baseline and after 6 months. At baseline patients will be randomized (2:1) to either an allogenic (from donors) infusion of collected feces (fecal microbiota transplantation, FMT) (or no procedure in case of allocation to placebo) in the duodenum-jejunum. The infusion will be performed through a standard nasojejunal tube, that will be placed during endoscopy. Infusion of feces will be performed at time 0 and repeated at month 6. The patients allocated to placebo arm will not receive treatment, but will undergo intestinal biopsy.

Upper GI endoscopy 12 months after FMT will be performed only to identify specific microbioma and mucosal immunological evaluation. Fecal samples and small intestine biopsy samples (at baseline, before treatment, and at month 6 and 12) will be obtained from patients to perform the gut microbiota typing.

Every endoscopic procedure will be performed with sedation of the patient. Feces for FMT will be obtained by healthy donors for C. difficile infection. Procedures that are usually performed for the selection of donors for transplantation of feces are as follows. Potential donors stool will be chosen in healthy volunteers that will have given a questionnaire with questions about lifestyle, health status, current therapy, etc., significant clinical symptoms of gastrointestinal disease, etc.. Based on this questionnaire, the potential donor will be considered eligible if excluded: I) Habits of life and risk behaviors, II) Concomitant significant known disorders, III) chronic or recent use of concomitant medications that may interfere with the state of the intestinal microflora (eg, antibiotics), IV) Clinical symptoms indicative of gastrointestinal disease or other diseases of importance, V) Personal or family medical history known of neurodegenerative diseases or other autoimmune diseases.

Moreover, each suitable potential donor will be subjected to the following screening tests: I) Examination of stool for Clostridium difficile bacterial pathogens and protozoa and helminths of the small intestine and colon, Vancomycin-resistant Enterococci (VRE ), Methicillin-resistant Staphylococcus aureus (MRSA), Gram-negative Multidrug-Resistant Organisms (MDR), II) Serological screening for hepatitis virus A,B and C, HIV 1-2, Treponema pallidum, H. pylori, blood count with differential, dose transaminasemia, creatinine and C-reactive protein.

Potential donors negative for this screening will be considered definitively suitable and will be invited to give a stool sample to prepare than for the fecal transplant. The donation will be made in the appropriate circles in the Department of Internal Medicine and Gastroenterology, and the preparation of faeces (manual homogenization in 500 mL of saline solution) for infusion will be performed at the Unit of Analysis 2 ° (Virology and Microbiology).

Analysis of T cell sub-populations will be performed both in peripheral blood and gut mucosa: especially the ratio T Regulatory cells (Tregs)/Th17 cells A Contract Research Organization (CRO) will be in charge for study monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a laboratory supported, clinically "probable" or "definite" amyotrophic lateral sclerosis according to the Revised El Escorial criteria (Brooks, 2000)
* Sporadic or familial ALS
* Female or male patients aged between 18 and 70 years old
* Disease duration from symptoms onset no longer than 18 months at the screening visit
* Patients treated with a stable dose of Riluzole (100 mg/day) for at least 30 days prior to screening
* Patients with a weight > 50 kg and a BMI ≥18
* Patients with a FVC (Forced Vital Capacity) equal or more than 70% predicted normal value for gender, height, and age at the screening visit
* Patients able and willing to comply with study procedures as per protocol
* Patients able to understand, and capable of providing informed consent at screening visit prior to any protocol-specific procedures
* Use of effective contraception both for males and females

Exclusion Criteria:

* Known organic gastrointestinal disease
* History of gastrointestinal malignancy; ongoing malignancies
* Use of immunosuppressive or chemotherapy within the past 2 years
* Celiac disease and/or food (e.g.lactose) intolerance
* Previous gastrointestinal surgery
* Any condition that would make endoscopic procedures contraindicated
* Acute infections requiring antibiotics
* Antimicrobial treatment or probiotics 4 weeks prior to screening
* Severe comorbidities (heart, renal, liver failure); severe renal (eGFR< 30ml/min/1.73m2), or liver failure or liver aminotransferase (ALT/AST > 2x Upper limit of normal),
* Autoimmune diseases, inflammatory disorders (SLE, Rheumatoid arthritis, connective tissue disorder) or chronic infections (HIV, hepatitis B or C infection)
* Abuse of alcohol or drugs
* HIV, tuberculosis, hepatitis
* Participation in clinical trials <30 days before screening
* Existing blood dyscrasia (e.g., myelodysplasia)
* White blood cells<4,000/mm³, platelets count<100,000/mm³, hematocrit<30%
* Patients who underwent non-invasive ventilation, tracheotomy and /or gastrostomy
* Women who are pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Tregs number | 6 months
  to assess whether FMT increases Tregs' number in ALS patients treated with FMT compared to the control arm

SECONDARY OUTCOMES:
Change in T cell subsets frequency in blood and gut tissue samples | 12 months (at time points: baseline, month 3 - 6 (both arms)- 9 -12 (both arms))
  Change from baseline to each time point (month 3, 6, 9, 12) of the T cell distribution especially the ratio Tregs/Th1 or Tregs/Th17comparing FMT arm and placebo arm.
Change in heavy neurofilaments levels in CSF | 6 months (at baseline and at month 6)
  assessment of ongoing disease activity by measuring neurofilaments in CSF only after a proper given consent (lumbar puncture will not be mandatory)
Changes in levels of pro-inflammatory cytokines and cytokines linked to T cell proliferation and differentiation | 6 months (at baseline and at month 6)
  Changes from baseline to each time point (month 3, 6, 9, 12) in inflammatory status (cytokines profile in CSF) comparing FMT and placebo arm, only after a proper given consent (lumbar puncture will not be mandatory). We will measure: MIP1a, IL-27, IL-1β, IL-2, IL-4, IL-5, IP-10, IL-6, IL-8, IL-10, IL-12p70, IL-13, IL-17A, IFNγ, GM-CSF, TNFα, IFNα, MCP-1, IL-9, P-selectin, IL-1α, IL-23, IL-18, IL-21, sICAM-1, IL-22, E-selectin content using specifically assembled kits (Custom Mix&Match panel Human Panel- 27 Plex) for Luminex Screening Assays (Affymetrix, eBioscience).
Changes in microbiota profile | 12 months (at baseline and at month 6 and 12)
  analysis of fecal, gut and saliva samples to assess whether FMT consistently modifies microbiota in treated patients versus placebo arm
Incidence of Adverse Events | 12 months ( at screening, baseline, month 1-3-6-7-9-12)
  Patients will be monitored with particular attention to possible side effects, including but not limited to increased risk of infections, constipation, diarrhea, pain, nausea, headache, fever. Routine blood samples will be performed at each neurological examination including blood cell count, serum cholesterol and triglycerides, liver and renal function, urine examination, fecal calprotectin.
Tracheostomy free survival | 12 months
  Overall survival from randomization to date of documented death or tracheostomy
Forced vital capacity (FVC) | 12 months (at baseline and month 3, 6, 9, 12)
  respiratory function
disease progression | 12 months (at baseline and month 3, 6, 9, 12)
  Amyotrophic lateral sclerosis functional rating scale-revised score, a scale which measures individual functioning through questions regarding communication, eating, motricity and respiration (values: maximum 48 corresponding to no disability; minimum 0 corresponding to extreme disability; higher values represent a good outcome)
quality of life: Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | 12 months (at baseline and month 6 and 12)
  measurement of quality of life by changes in Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) a scale used to measure the subjective well-being of patients with amyotrophic lateral sclerosis; it includes 40 items / questions. Dimension scores are coded on a scale of 0 (perfect health as assessed by the measure) to 100 (worst health as assessed by the measure).

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Clinica Neurologica, Ospedale Clinicizzato "SS Annunziata", Chieti
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - UO Neurofisiopatologia, Azienda Ospedaliera dì Perugia, Perugia
  - Catholic University of Sacred Heart - Fondazione Policlinico "A. Gemelli", Roma
  - NEuroMuscular Omnicentre Centre (NeMO), Fondazione Serena Onlus-Fondazione Policlinico A. Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data will be made available after study completion upon specific request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available at study completion (after final data analysis)
Access Criteria: specific personal request by the subject

REFERENCES:
- [Result] ALSUntangled Group. ALS Untangled No. 21: Fecal transplants. Amyotroph Lateral Scler Frontotemporal Degener. 2013 Sep;14(5-6):482-5. doi: 10.3109/21678421.2013.814981. Epub 2013 Jul 22. No abstract available. PMID 23870000
- [Result] Amedei A, Della Bella C, Niccolai E, Stanflin N, Benagiano M, Duranti R, Del Prete G, Murphy TF, D'Elios MM. Moraxella catarrhalis-specific Th1 cells in BAL fluids of chronic obstructive pulmonary disease patients. Int J Immunopathol Pharmacol. 2009 Oct-Dec;22(4):979-90. doi: 10.1177/039463200902200413. PMID 20074461
- [Result] Backhed F, Ley RE, Sonnenburg JL, Peterson DA, Gordon JI. Host-bacterial mutualism in the human intestine. Science. 2005 Mar 25;307(5717):1915-20. doi: 10.1126/science.1104816. PMID 15790844
- [Result] Baxter M, Colville A. Adverse events in faecal microbiota transplant: a review of the literature. J Hosp Infect. 2016 Feb;92(2):117-27. doi: 10.1016/j.jhin.2015.10.024. Epub 2015 Dec 15. PMID 26803556
- [Result] Beers DR, Henkel JS, Zhao W, Wang J, Huang A, Wen S, Liao B, Appel SH. Endogenous regulatory T lymphocytes ameliorate amyotrophic lateral sclerosis in mice and correlate with disease progression in patients with amyotrophic lateral sclerosis. Brain. 2011 May;134(Pt 5):1293-314. doi: 10.1093/brain/awr074. PMID 21596768
- [Result] Bienenstock J, Kunze W, Forsythe P. Microbiota and the gut-brain axis. Nutr Rev. 2015 Aug;73 Suppl 1:28-31. doi: 10.1093/nutrit/nuv019. PMID 26175487
- [Result] Boillee S, Yamanaka K, Lobsiger CS, Copeland NG, Jenkins NA, Kassiotis G, Kollias G, Cleveland DW. Onset and progression in inherited ALS determined by motor neurons and microglia. Science. 2006 Jun 2;312(5778):1389-92. doi: 10.1126/science.1123511. PMID 16741123
- [Result] Borody TJ, Khoruts A. Fecal microbiota transplantation and emerging applications. Nat Rev Gastroenterol Hepatol. 2011 Dec 20;9(2):88-96. doi: 10.1038/nrgastro.2011.244. PMID 22183182
- [Result] Bradley WG, Borenstein AR, Nelson LM, Codd GA, Rosen BH, Stommel EW, Cox PA. Is exposure to cyanobacteria an environmental risk factor for amyotrophic lateral sclerosis and other neurodegenerative diseases? Amyotroph Lateral Scler Frontotemporal Degener. 2013 Sep;14(5-6):325-33. doi: 10.3109/21678421.2012.750364. Epub 2013 Jan 4. PMID 23286757
- [Result] Brandt LJ. Fecal Microbiota Transplant: Respice, Adspice, Prospice. J Clin Gastroenterol. 2015 Nov-Dec;49 Suppl 1:S65-8. doi: 10.1097/MCG.0000000000000346. PMID 26447968
- [Result] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Result] Erny D, Hrabe de Angelis AL, Jaitin D, Wieghofer P, Staszewski O, David E, Keren-Shaul H, Mahlakoiv T, Jakobshagen K, Buch T, Schwierzeck V, Utermohlen O, Chun E, Garrett WS, McCoy KD, Diefenbach A, Staeheli P, Stecher B, Amit I, Prinz M. Host microbiota constantly control maturation and function of microglia in the CNS. Nat Neurosci. 2015 Jul;18(7):965-77. doi: 10.1038/nn.4030. Epub 2015 Jun 1. PMID 26030851
- [Result] Frank DN, St Amand AL, Feldman RA, Boedeker EC, Harpaz N, Pace NR. Molecular-phylogenetic characterization of microbial community imbalances in human inflammatory bowel diseases. Proc Natl Acad Sci U S A. 2007 Aug 21;104(34):13780-5. doi: 10.1073/pnas.0706625104. Epub 2007 Aug 15. PMID 17699621
- [Result] Hardiman O, van den Berg LH. Edaravone: a new treatment for ALS on the horizon? Lancet Neurol. 2017 Jul;16(7):490-491. doi: 10.1016/S1474-4422(17)30163-1. Epub 2017 May 15. No abstract available. PMID 28522180
- [Result] Henkel JS, Beers DR, Wen S, Rivera AL, Toennis KM, Appel JE, Zhao W, Moore DH, Powell SZ, Appel SH. Regulatory T-lymphocytes mediate amyotrophic lateral sclerosis progression and survival. EMBO Mol Med. 2013 Jan;5(1):64-79. doi: 10.1002/emmm.201201544. Epub 2012 Nov 9. PMID 23143995
- [Result] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Result] Khanna S. Microbiota Replacement Therapies: Innovation in Gastrointestinal Care. Clin Pharmacol Ther. 2018 Jan;103(1):102-111. doi: 10.1002/cpt.923. Epub 2017 Nov 14. PMID 29071710
- [Result] Kimura F, Fujimura C, Ishida S, Nakajima H, Furutama D, Uehara H, Shinoda K, Sugino M, Hanafusa T. Progression rate of ALSFRS-R at time of diagnosis predicts survival time in ALS. Neurology. 2006 Jan 24;66(2):265-7. doi: 10.1212/01.wnl.0000194316.91908.8a. PMID 16434671
- [Result] Kadowaki A, Miyake S, Saga R, Chiba A, Mochizuki H, Yamamura T. Gut environment-induced intraepithelial autoreactive CD4(+) T cells suppress central nervous system autoimmunity via LAG-3. Nat Commun. 2016 May 20;7:11639. doi: 10.1038/ncomms11639. PMID 27198196
- [Result] Lee YK, Menezes JS, Umesaki Y, Mazmanian SK. Proinflammatory T-cell responses to gut microbiota promote experimental autoimmune encephalomyelitis. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4615-22. doi: 10.1073/pnas.1000082107. Epub 2010 Jul 26. PMID 20660719
- [Result] Longstreth WT Jr, Meschke JS, Davidson SK, Smoot LM, Smoot JC, Koepsell TD. Hypothesis: a motor neuron toxin produced by a clostridial species residing in gut causes ALS. Med Hypotheses. 2005;64(6):1153-6. doi: 10.1016/j.mehy.2004.07.041. PMID 15823706
- [Result] Mayer EA, Tillisch K, Gupta A. Gut/brain axis and the microbiota. J Clin Invest. 2015 Mar 2;125(3):926-38. doi: 10.1172/JCI76304. Epub 2015 Feb 17. PMID 25689247
- [Result] Moreno-Igoa M, Calvo AC, Penas C, Manzano R, Olivan S, Munoz MJ, Mancuso R, Zaragoza P, Aguilera J, Navarro X, Osta Pinzolas R. Fragment C of tetanus toxin, more than a carrier. Novel perspectives in non-viral ALS gene therapy. J Mol Med (Berl). 2010 Mar;88(3):297-308. doi: 10.1007/s00109-009-0556-y. PMID 19921501
- [Result] Piccione EA, Sletten DM, Staff NP, Low PA. Autonomic system and amyotrophic lateral sclerosis. Muscle Nerve. 2015 May;51(5):676-9. doi: 10.1002/mus.24457. Epub 2015 Mar 31. PMID 25211238
- [Result] Round JL, Mazmanian SK. Inducible Foxp3+ regulatory T-cell development by a commensal bacterium of the intestinal microbiota. Proc Natl Acad Sci U S A. 2010 Jul 6;107(27):12204-9. doi: 10.1073/pnas.0909122107. Epub 2010 Jun 21. PMID 20566854
- [Result] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Result] Tremlett H, Bauer KC, Appel-Cresswell S, Finlay BB, Waubant E. The gut microbiome in human neurological disease: A review. Ann Neurol. 2017 Mar;81(3):369-382. doi: 10.1002/ana.24901. Epub 2017 Mar 20. PMID 28220542
- [Result] van Es MA, Hardiman O, Chio A, Al-Chalabi A, Pasterkamp RJ, Veldink JH, van den Berg LH. Amyotrophic lateral sclerosis. Lancet. 2017 Nov 4;390(10107):2084-2098. doi: 10.1016/S0140-6736(17)31287-4. Epub 2017 May 25. PMID 28552366
- [Result] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Result] Wang S, Xu M, Wang W, Cao X, Piao M, Khan S, Yan F, Cao H, Wang B. Systematic Review: Adverse Events of Fecal Microbiota Transplantation. PLoS One. 2016 Aug 16;11(8):e0161174. doi: 10.1371/journal.pone.0161174. eCollection 2016. PMID 27529553
- [Result] Wu S, Yi J, Zhang YG, Zhou J, Sun J. Leaky intestine and impaired microbiome in an amyotrophic lateral sclerosis mouse model. Physiol Rep. 2015 Apr;3(4):e12356. doi: 10.14814/phy2.12356. PMID 25847918
- [Result] Zhao W, Xie W, Xiao Q, Beers DR, Appel SH. Protective effects of an anti-inflammatory cytokine, interleukin-4, on motoneuron toxicity induced by activated microglia. J Neurochem. 2006 Nov;99(4):1176-87. doi: 10.1111/j.1471-4159.2006.04172.x. Epub 2006 Oct 2. PMID 17018025